CLINICAL TRIAL: NCT01981798
Title: The Long-term Effect of an Outpatient Intervention Program With a Behavioral Therapy Approach in Patients With Chronic Back or Neck Pain With a Focus on Psychosocial Aspects
Brief Title: Effect of an Outpatient Intervention Program in Patients With Chronic Back or Neck Pain
Acronym: CPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Orthopedic Hospital Vienna Speising (Other)
Responsible Party: Principal Investigator, Florian Wepner, Dr., Orthopedic Hospital Vienna Speising
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Praev123
Record Dates: First submitted 2013-08-29; First posted 2013-11-13 (Estimated); Last update posted 2013-11-13 (Estimated); Status verified 2013-11

CONDITIONS: Chronic Low Back Pain; Neck Pain
Keywords: outpatient intervention program; behavioral therapy approach; unspecific back pain; unspecific neck pain; chronic pain; physiotherapy; occupational therapy; psychosocial aspects; fear avoidance beliefs; health-related quality of life
MeSH Terms: conditions — Neck Pain; Chronic Pain | interventions — Physical Therapy Modalities; Occupational Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Training group (Active Comparator): Physiotherapy and occupational therapy: Training group received 9 units of physiotherapy and 2 units of occupational therapy, each with a duration of one hour.
  Interventions: Behavioral: Physiotherapy and occupational therapy
- Control Group (No Intervention): Members of the control group were referred to their general practitioner or specialist for further care.

INTERVENTIONS:
Behavioral: Physiotherapy and occupational therapy — Members of the training group received 9 units of physiotherapy and 2 units of occupational therapy, each with a duration of one hour. Every patient of the IG was trained to perform a neck or back intervention program specifically suited to his/her needs. The training was conducted in a single session by one of three experienced physiotherapists (with mean work experience of 6 years). After this training the patients completed eight group training units consisting a maximum number of 8 participants, each unit with a duration of one hour, over a maximum period of six weeks.
  Arms: Training group

SUMMARY:
To investigated whether an ambulant intervention program with a behavioral therapy approach would exert a long-term effect on chronic unspecific back or neck pain. Specifically, the effect on patients with pronounced fear avoidance behavior and/or with psychosocial limitations was addressed.

DETAILED DESCRIPTION:
BACKGROUND: Sustained success of ambulant intervention programs consisting of individual and group physiotherapy in patients with with chronic unspecific back or neck pain (cBP) has not been conclusively proven. It's still not clear whether one can achieve such success by devoting greater attention to psychosocial factors.

OBJECTIVE: We investigated whether an ambulant intervention program with a behavioral therapy approach would exert a long-term effect on cBP. Specifically, the effect on patients with pronounced fear avoidance behavior and/or with psychosocial limitations was addressed.

DESIGN: Prospective, randomized controlled trial

SETTINGS, INTERVENTION: 64 patients were assigned to intervention group (IG) and 57 to control group (CG). All were examined, informed about cBP, and were encouraged to stay active and perform exercises according to specific instructions provided in a neck- or back-book. The IG received 9 units of physiotherapy and 2 units of occupational therapy, conducted with a behavioral therapy approach. Efficacy of treatment was evaluated after 6 and 58 weeks.

MEASUREMENTS: Pain (VAS), quantity of painkillers consumed, sick leave days, Oswestry-Disability-Index (ODI), SF-36, FABQ.

ELIGIBILITY:
Inclusion Criteria:

* minimum age 18 years, maximum age: men 55 years, women 50 years.
* the patients had been on sick leave for a minimum of 4 and a maximum of 22 days during the preceding 12 months because of nonspecific spinal symptoms in the back or neck.
* The patients had to be working at the start of the study.

Exclusion Criteria:

* Specific causes of spinal symptoms (after spinal surgery, known vertebral body fractures, disk prolapse with motor deficits or other radicular lesions, tumor, osteomyelitis, spondylodiscitis, rheumatic disease, osteoporosis).
* Retired persons, those in the process of being screened for retirement, unemployed persons,
* pregnancy or persons on maternity leave
* Planned surgery during the phase of intervention
* persons who were unable to participate in the intervention program for other reasons (physical, psychological, linguistic or organizational).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 121 (Actual)
Dates: Start 2006-03; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Pain | After 0 / 6 / 58 Weeks
  To evaluate the main hypothesis, current pain and mean pain during the preceding week and the preceding 3 months were determined on a visual analog scale (VAS; 0-100, lower scores indicate less severe pain)

SECONDARY OUTCOMES:
Social function, psychological wellbeing and emotional role function | After 0 / 6 / 58 weeks
  To evaluate social function, psychological wellbeing and emotional role function we used the 36-item short form health survey (SF-36; scales 0-100, lower scores indicate poorer social, psychological and emotional quality of life)
Functional impairment | After 0 / 6 / 58 weeks
  The Oswestry disability index was used to measure functional impairment.
Anxiety, insecurity in social contacts and compulsiveness | After 0 / 6 / 58 weeks
  Anxiety, insecurity in social contacts and compulsiveness were registered on the brief symptoms inventory (BSI), which is an abridged version of SCL-90_R. The BSI addresses subjective experience of impairment based on a list of symptoms that are partly physical and partly psychological. The time frame is seven days.
Sick leave days | After 0 / 58 weeks
  The number of (self-reported) days of sick leave due to pain during the preceding twelve months were inquired.
Painkillers | After 0 / 58 weeks
  The number of painkillers taken per day were inquired.
Fear avoidance behavior | After 0 / 6 / 58 weeks
  Fear avoidance behavior was determined by means of the fear avoidance beliefs questionnaire (FABQ; scale 0-66; lower scores indicate lower fear-avoidance beliefs)

CONTACTS AND LOCATIONS:
Overall Officials: Florian Wepner, Dr., Principal Investigator — Orthopedic Hospital Vienna Speising; Martin Friedrich, Prof., Study Chair — Orthopedic Hospital Vienna Speising; Julia Hahne, Mag., Study Director — Orthopedic Hospital Vienna Speising
Locations (1):
- Orthopedic Hospital Vienna Speising, Vienna, Vienna, Austria

REFERENCES:
- [Background] Chou R, Loeser JD, Owens DK, Rosenquist RW, Atlas SJ, Baisden J, Carragee EJ, Grabois M, Murphy DR, Resnick DK, Stanos SP, Shaffer WO, Wall EM; American Pain Society Low Back Pain Guideline Panel. Interventional therapies, surgery, and interdisciplinary rehabilitation for low back pain: an evidence-based clinical practice guideline from the American Pain Society. Spine (Phila Pa 1976). 2009 May 1;34(10):1066-77. doi: 10.1097/BRS.0b013e3181a1390d. PMID 19363457
- [Background] Airaksinen O, Brox JI, Cedraschi C, Hildebrandt J, Klaber-Moffett J, Kovacs F, Mannion AF, Reis S, Staal JB, Ursin H, Zanoli G; COST B13 Working Group on Guidelines for Chronic Low Back Pain. Chapter 4. European guidelines for the management of chronic nonspecific low back pain. Eur Spine J. 2006 Mar;15 Suppl 2(Suppl 2):S192-300. doi: 10.1007/s00586-006-1072-1. No abstract available. PMID 16550448
- [Background] Waddell G, Newton M, Henderson I, Somerville D, Main CJ. A Fear-Avoidance Beliefs Questionnaire (FABQ) and the role of fear-avoidance beliefs in chronic low back pain and disability. Pain. 1993 Feb;52(2):157-168. doi: 10.1016/0304-3959(93)90127-B. PMID 8455963
- [Background] Klenerman L, Slade PD, Stanley IM, Pennie B, Reilly JP, Atchison LE, Troup JD, Rose MJ. The prediction of chronicity in patients with an acute attack of low back pain in a general practice setting. Spine (Phila Pa 1976). 1995 Feb 15;20(4):478-84. doi: 10.1097/00007632-199502001-00012. PMID 7747233
- [Background] van Middelkoop M, Rubinstein SM, Kuijpers T, Verhagen AP, Ostelo R, Koes BW, van Tulder MW. A systematic review on the effectiveness of physical and rehabilitation interventions for chronic non-specific low back pain. Eur Spine J. 2011 Jan;20(1):19-39. doi: 10.1007/s00586-010-1518-3. Epub 2010 Jul 18. PMID 20640863
- [Background] Somerville S, Hay E, Lewis M, Barber J, van der Windt D, Hill J, Sowden G. Content and outcome of usual primary care for back pain: a systematic review. Br J Gen Pract. 2008 Nov;58(556):790-7, i-vi. doi: 10.3399/bjgp08X319909. PMID 19000402
- [Background] Burton AK, Waddell G, Tillotson KM, Summerton N. Information and advice to patients with back pain can have a positive effect. A randomized controlled trial of a novel educational booklet in primary care. Spine (Phila Pa 1976). 1999 Dec 1;24(23):2484-91. doi: 10.1097/00007632-199912010-00010. PMID 10626311
- [Background] Hides JA, Jull GA, Richardson CA. Long-term effects of specific stabilizing exercises for first-episode low back pain. Spine (Phila Pa 1976). 2001 Jun 1;26(11):E243-8. doi: 10.1097/00007632-200106010-00004. PMID 11389408
- [Background] Lamb SE, Hansen Z, Lall R, Castelnuovo E, Withers EJ, Nichols V, Potter R, Underwood MR; Back Skills Training Trial investigators. Group cognitive behavioural treatment for low-back pain in primary care: a randomised controlled trial and cost-effectiveness analysis. Lancet. 2010 Mar 13;375(9718):916-23. doi: 10.1016/S0140-6736(09)62164-4. Epub 2010 Feb 25. PMID 20189241
- [Background] Johnson RE, Jones GT, Wiles NJ, Chaddock C, Potter RG, Roberts C, Symmons DP, Watson PJ, Torgerson DJ, Macfarlane GJ. Active exercise, education, and cognitive behavioral therapy for persistent disabling low back pain: a randomized controlled trial. Spine (Phila Pa 1976). 2007 Jul 1;32(15):1578-85. doi: 10.1097/BRS.0b013e318074f890. PMID 17621203